# ORthopaedic trauma Anemia with Conservative versus Liberal transfusion (ORACL) (NCT02972593)

Brian Mullis, MD
Chief, Orthopaedic Trauma Service
Eskenazi Health, Fifth Third Bank Building
720 Eskenazi Avenue
2<sup>nd</sup> Floor, Suite 2-S
Indianapolis, IN 46202
Associate Professor
Indiana University School of Medicine
Assistant: 317-880-3600

Office: 317-880-3591 Fax: 317-880-0138

#### **Participating Sites:**

Eskenazi Hospital-Orthopaedics (Site PI: Karl Shively, MD)
Methodist Hospital-Orthopaedics (Site PI: Walter Virkus, MD)
WellStar Atlanta Medical Center (Site PI: Jennifer Bruggers, MD)
Atrium Health Musculoskeletal Institute-Charlotte, NC (Site PI: Laurence Kempton, MD)

#### **Table of Contents:**

#### **Study Schema**

- 1.0 Background
- 2.0 Rationale and Specific Aims
- 3.0 Inclusion/Exclusion Criteria
- 4.0 Enrollment/Randomization
- 5.0 Study Procedures
- 6.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others
- 7.0 Study Withdrawal/Discontinuation
- **8.0** Statistical Considerations
- 9.0 Privacy/Confidentiality Issues
- 10.0 Follow-up and Record Retention
- 11.0 Investigator Environment and Support
- 12.0 References

**Appendix A: Screening Form CRF** 

**Appendix B: Contact Information CRF** 

**Appendix C: Pre-injury MFA CRF** 

**Appendix D: Follow-up MFA CRF** 

**Appendix E: 2 minute walk test CRF** 

**Appendix F: Adverse Event CRF** 

**Appendix G: Protocol Deviation CRF** 

Appendix H: Escape Criteria CRF

**Appendix I: Length of Hospital Stay CRF** 

Appendix J: AAOS Abstract February 2011

Appendix K: American Journal of Orthopaedics Article, 2015

#### 1.0 Background

Over 13 million units of blood are transfused each year. While transfusion can certainly be life saving, numerous studies over the last twenty years have shown significant, dose-dependent increases in morbidity, mortality, and cost with each unit of packed red blood cells transfused. {Leal-Noval, 2001 #1} Transfusion is one of the most common interventions made in the critically ill population, however the negative effects of transfusion-related infection is well documented in recent literature. {Leal-Noval, 2001 #1;Leal-Noval, 2001 #1;Hebert, 1999 #2;Carson, 1999 #3;Edna, 1992 #6;Hill, 2003 #8;Vincent, 2002 #9;Taylor, 2002 #10} There is no question that transfusion of blood products can be life-saving to an acutely ill trauma patient, but there is little evidence to help the Orthopaedic Surgeon decide when a transfusion is indicated in an asymptomatic anemic patient who is no longer in need of acute resuscitation.

Several studies have analyzed healthy individuals with an isovolemic reduction in hemoglobin to a level of 5.0 (g/dL). {Leung, 2000 #16; Weiskopf, 1998 #17} They found no significant compromise in oxygen delivery to the tissues. Currently there is a lack of clinical data to suggest adequate red blood cell (RBC) transfusion endpoints in trauma surgery. {Johnston, 2006 #18} Given the lack of evidence to support transfusion triggers for young, healthy, asymptomatic Orthopaedic trauma patients, the purpose of this study will be to investigate the risk of complications associated with permissive anemia in this population.

Orthopaedic trauma patients treated at Eskenazi (previously Wishard) Hospital, a level 1 trauma center, are routinely allowed to be permissively anemic, or allowed to run as low as a Hemoglobin of 5 g/dL if they are young and healthy (see inclusion/exclusion criteria for objective definition) and asymptomatic from anemia. A retrospective review was performed using the inclusion/exclusion criteria proposed in this study to evaluate if a prospective study would be ethical and to provide a power analysis for number of patients needed to reject the null hypothesis. Over a 3 year period (2006-2009), 104 patients were identified who met the inclusion/exclusion criteria proposed in this study and were available for 1 year follow-up. This study controlled for Injury Severity Score, patient age, gender, and whether the patient had received multiple surgeries. We found that patients who were allowed to be permissively anemic (allowed to drop to a Hgb of 5 g/dL if asymptomatic at rest) had a lower complication rate (p<0.01) than those who were transfused to maintain a higher hemoglobin. Additionally, there appeared to be a dosedependent affect (p=0.02) with higher complications seen in patients receiving multiple units of allogeneic blood. This data was presented at both the American Academy of Orthopaedic Surgery (2011) and Orthopaedic Trauma Association (2011) annual meetings and the manuscript is currently being reviewed for publication. This retrospective study does not prove causation of higher complication rates associated directly with transfusion, but does suggest there may be a lower complication rate in patients allowed to be permissively anemic. The largest barrier to publication of this retrospective study has been the repeated comments by reviewers that a prospective study is needed.

Dr. Mullis, Chief of Orthopaedic Trauma at Eskenazi Hospital, has met with the Chief of Anesthesia at Eskenazi Hospital, John Hasewinkel, and the Chief of Trauma for General Surgery, Gerry Gomez, to develop the inclusion and exclusion criteria listed

below so that this study might be completed in a multi-disciplinary approach with all providers agreeing to the inclusion and exclusion criteria and escape criteria listed below.

#### 2.0 Rationale and Specific Aims

Transfusion of Orthopaedic trauma patients is routinely done in asymptomatic individuals as there is no accepted national standard or recommendations from the American Academy of Orthopaedic Surgeons or the Orthopaedic Trauma Association for what level of anemia is appropriate in an asymptomatic patient. Individual practitioners typically make this decision based on anecdotal experiences and expert opinion. No prospective study has been performed to date to answer this question in this patient population.

The null hypothesis of this proposed pilot study is that no difference will be seen with a liberal transfusion strategy to keep a patient's hemoglobin above 7 g/dL versus a conservative strategy to keep the patient's hemoglobin above 5.5 g/dL in patients asymptomatic at rest. The primary outcome of this pilot study will be infection; defined as postoperative wound infection (superficial or deep) or other perioperative infection but not surgical site (urinary tract infection or pneumonia). Deep infection is defined as the need for intravenous antibiotics or a return to surgery for debridement. Superficial infection is defined as the use of oral antibiotics only successfully treat a surgical site infection. Secondary outcomes will include pulmonary embolism, deep venous thrombosis, acute renal failure or insufficiency, nonunion, delayed union, compartment syndrome, osteomyelitis, nerve palsy, anoxic brain injury, cardiac ischemia or infarct, pancreatitis, or death, and the musculoskeletal functional assessment. These same outcomes were evaluated in the retrospective study done at this institution which found no difference within any one complication, but when all complications were pooled there was a higher complication associated with the liberal transfusion strategy.

#### 3.0 Inclusion/Exclusion Criteria

#### Inclusion criteria:

- Trauma patients admitted to participating hospital with any Orthopaedic injury who have been determined to be stable by the Trauma Service (General Surgery) and are no longer within the resuscitation phase of initial treatment. This is defined as a normal urine output (greater than 0.5 ml/kg/hr) and a systolic blood pressure greater than 90 mmHg for greater than 6 hours without fluid bolus or transfusion during that time
- Age 18-50
- Hemoglobin less than 9 g/dL or expected drop below 9 g/dL with planned surgery

#### Exclusion criteria:

- Pregnant ( urine pregnancy test will be done as standard of care)
- Prisoner
- Head injury (Glasgow Coma Scale less than 8 over 48 hours from presentation)
- Known cardiac (coronary artery disease, atrial fibrillation, stent placement, congestive heart failure), renal (acute or chronic renal insufficiency or failure,

defined as having Serum Creatinine >1.2 at time of enrollment), liver (Childs C cirrhosis) or pulmonary disease (chronic obstructive pulmonary disease, abnormal pulmonary function tests or history of poor pulmonary function from any cause including acute traumatic conditions such as ARDS)

- Unlikely to follow up in the surgeon's estimation
- Sickle Cell Anemia
- History of cancer
- Preexisting weakness, paresthesias, deformities, or other conditions which might affect functional outcome in the surgeon's opinion
- Spinal cord injury
- Patients with burns expected to require operative treatment
- COVID positive

#### 4.0 Enrollment/Randomization

A consensus opinion was reached in a multidisciplinary manner with multiple members of the Trauma team (General Surgery), Anesthesia, Physical Medicine and Rehab, and the Orthopaedic Trauma Service. This team consisted of members from General Surgery (Timothy Hayward, Erik Streib, Clark Simons, Gerry Gomez), Anesthesia (John Hasewinkel, Jim Mitchell, Leilani Mullis), and Physical Medicine and Rehab (Angela Carbone) along with all members of the Orthopaedic Trauma Service (Jeff Anglen, Janos Ertl, Karl Shively) and the PI (Brian Mullis). The opinions in escape criteria and definitions will be referred to below as "consensus opinion". A biostatistician was consulted after he had reviewed the data from the retrospective study previously performed at this institution to help design an appropriately powered prospective randomized pilot study.

All Orthopaedic Trauma patients admitted to participating hospital will be screened for inclusion and exclusion criteria after they have been resuscitated and stabilized. The consensus opinion of the "stable" patient was defined as an awake and alert patient with normal urine output and systolic blood pressure greater than 90 mmHG for greater than 6 hours without fluid bolus or resuscitation. If a patient meets criteria for the study as noted above and is stable as defined above, the patient would be approached by either the Principal Investigator (PI) or a co-PI to determine interest and informed consent would be obtained for participation in the study. Patients who either refuse or are unable to consent will be tracked using the screening form. Enrollment would be performed in patients with a Hgb of 9 g/dL or less or in patients expected to drop below 9 g/dL with planned procedures or continued (controlled) bleeding. Randomization would not occur until the patient's Hgb dropped below 7 g/dL at which time a sealed envelope would be opened to determine if the patient would be randomized to a liberal transfusion strategy (transfuse to keep Hgb >7 g/dL) or a conservative strategy (transfuse to keep Hgb > 5.5 g/dL). If the patient's Hgb does not drop below 7.0 g/dL, randomization will not be done. Prior to starting enrollment, envelopes will be made by blinded personnel using a randomization list generated to assign subjects to receive treatment either after hemoglobin drops below 5.5 or after hemoglobin drops below 7.0. Randomization was

done with a block size of 4 to ensure the treatment allocation was balanced throughout the study recruitment period. Escape criteria have been established by the consensus group to allow transfusion in patients with clinical concerns for symptomatic or dangerous levels of anemia despite randomization arm (please see Escape Criteria outlined in section 5.0)

#### 5.0 Study Procedures

If the patient remains asymptomatic at rest (defined as no chest pain, shortness of breath, or dizziness), transfusion would be determined by randomization to the liberal transfusion strategy to maintain Hgb at 7 g/dL or the conservative transfusion strategy of 5.5 g/dL. After each unit of blood is transfused a Hgb level would be checked to ensure appropriate Hgb levels are maintained as well as routine clinical practice (typically daily Hgb levels drawn until at least 2 consecutive days show no further drop with no further procedures or bleeding expected). If the patient's Hgb does not drop below 7.0 g/dL, randomization will not be done but patient will still be followed and patient outcomes will be collected as part of a non-treatment group.

As noted in Section 4.0, a consensus group consisting of multiple physicians and the service chiefs from the Trauma Service (General Surgery), Orthopaedic Trauma Service, Anesthesia, and Physical Medicine and Rehab agreed to the following escape criteria to transfuse regardless of Hgb level or arm of randomization:

#### Escape Criteria

- 1. Patient has any of the following symptoms at rest: chest pain, shortness of breath, dizziness
- 2. Patient has a mean arterial pressure less than 50 mmHg that is not responsive to fluid resuscitation
- 3. At any time the patient's heart rate increases by more than 30% above baseline while under anesthesia
- 4. The patient's urine output drops to less than 0.5 mL/kg/hour and remains decreased despite adequate rehydration with fluids
- 5. Any objective evidence of cardiac ischemia including the following: EKG changes such as ST depression, an elevation of serum cardiac markers, a base deficit greater than 6, lactate greater than 2.5 that does not respond to fluid resuscitation
- 6. A decrease in systolic blood pressure by 10% or more with exercise (physical therapy) that does not improve with fluid resuscitation
- 7. Uncontrolled source of hemorrhage

In addition to being followed daily while inpatient, patients would be followed at routine intervals following injury: 2 weeks, 6 weeks, 3 months, 6 months, 9 months, and 1 year. Radiographic and clinical data will be collected specific to the patient's musculoskeletal injury and based on standard of care. The primary outcome is infection defined as superficial infection (cellulitis treated with oral antibiotics) or deep infection (requires IV antibiotics or surgical debridement), osteomyelitis, pneumonia, urinary tract infection.

Secondary outcomes include renal insufficiency, cardiac ischemia or myocardial infarction, deep venous thrombosis, or any other medical complication encountered in the patient's hospital or post-discharge course felt to be possibly related to the patient's injury, procedure, or as a result of transfusion. Secondary outcomes will also include standardized patient outcome scores; specifically, the Musculoskeletal Functional Assessment (MFA) done at baseline, 6 months, and 1 year, and the two minute walk test which would be conducted daily by a certified physical therapist while the patient is an inpatient and after they have been cleared for ambulation. Length of hospital stay will be recorded. Return to surgery or repeat hospitalization due to a complication will be other secondary outcomes. Completion of the Musculoskeletal Functional Assessment at 6 months and 1 year may be done via phone or mail, if the subject is unable or unwilling to return for clinic follow up.

Other possible risks, no matter which group subjects are randomized to, are:

- Infection
- Osteomyelitis
- Pneumonia
- Urinary tract infection
- Renal insufficiency
- Acute renal failure
- Cardiac ischemia or infarct
- Myocardial infarction
- Pancreatitis
- Deep venous thrombosis
- Pulmonary embolism
- Anoxic brain injury
- Death
- Delayed union
- Non-union
- Compartment syndrome
- Nerve palsy

Risk level is the same for all events listed. These risks are possible but there is a low chance for occurrence.

## 6.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others

Any adverse event identified by a member of the care or research team from any participating site will be documented in writing and the lead site principal investigator will be notified of adverse events as they occur. All serious adverse events, protocol deviations, and noncompliance will be reported to the IRB in accordance with IU IRB policies and procedures. Significant adverse events that meet the policy criteria will be reported to the IRB as they occur. All other adverse events will be documented and reported to the IRB at time of continuing review.

A Data Safety Monitoring Plan (DSMP) will be in place to compare provisional outcomes prior to final enrollment. Per the DSMP, an orthopaedic surgeon not involved with the study will serve as the reviewer, looking at study data for obvious trends in higher complications in one study group. Monitoring of data that has been collected from all participating sites will be done every 6 months and findings will be submitted to the IRB at the time of continuing review. The data safety monitoring board will be comprised of: Todd McKinley-Independent Orthopaedic Surgeon, practices at Methodist (Board Chair), Dana Brock-Anesthesiologist at Eskenazi, Clark Simons-General Surgeon at Eskenazi, and Colin Terry- Biostatistician at Methodist. Qing Yu, PhD- Assistant Research Professor of Orthopaedic Surgery at IU will provide statistical analysis as needed. The DSMB has the independent ability to stop the study at any time if there is a concern for patient safety.

#### 7.0 Study Withdrawal/Discontinuation

Subjects have the right to withdraw from the study at any time and for any reason without prejudice to future medical care. If a subject wishes to withdraw from the study, they must notify a member of the research team. Once withdrawn, no further data will be collected from the subject.

#### 8.0 Statistical Considerations

#### Sample size:

This is a pilot study since the primary purpose of this study is to collect preliminary data on estimating the complication rates for orthopedic trauma patients who will receive blood transfusion either with a liberal transfusion strategy or a conservative strategy. The primary outcome of this study is whether a patient develops a complication while following a

conservative or liberal transfusion strategy for anemia. From our retrospective study, we anticipate the true complication rate would be anywhere between 30% and 50%. We want to estimate this proportion with 95% confidence and no more than 14% margin of error. With a sample size of 50 per group we would able to reach this goal. For example, if the true proportion is 40%, the margin of error will be 13.6% and the maximum margin of error would be 13.9% when the true proportion is 50%.

Up to 370 subjects will be enrolled as part of the non-treatment group.

#### Data Analysis:

The primary endpoint is a dichotomous outcome, the presence or absence of a complication at post blood transfusion. A point estimate (sample proportion) and a 95% confidence interval for the proportion will be reported. This proportion will be computed for each of the two blood transfusion strategies. Although we did not power the study to detect a difference in complication rate between two strategies, we will compare the complication rates between two groups of patients. Descriptive statistics, like, mean, median, standard deviation for continuous outcomes will be used to describe the subjects' characteristics at baseline. Frequency counts and percent will be used for the categorical outcomes. Baseline clinical and demographic data will be compared between two groups to assess the effectiveness of the randomization. Dichotomous and ordinal variables will be examined using chi-square tests and continuous measures with Student's t-tests. Exploratory analysis will be performed to compute p-values which will be presented as an aid to evaluate the overall comparability of the treatment groups at baseline. Logistic regression model will be used to compare the complication rate or infection rate between two groups and baseline covariates will be included in the model if two groups are found to be significantly different in those covariates.

#### 9.0 Privacy/Confidentiality Issues

Standard HIPAA practices will apply to all sensitive data recorded for study purposes. All attempts will be made to maintain confidentiality between study participants and the research team. Computer/files will be password protected, kept behind locked doors, and located in an area with no public access.

#### 10.0 Follow-up and Record Retention

Duration of the study will last approximately 3 years or until 100 patients have been enrolled with one year follow-up and all necessary data has been collected and analyzed.

Upon study completion, records will be retained for a minimum of 7 years as required by state law. After mandatory retention period, sensitive information will be disposed of by means of hospital provided secure document disposal.

#### 11.0 Investigator Environment and Support

The Orthopaedic research team based at Eskenazi Health has a long history of successful participation in prospective trauma research studies. The PI has successfully partnered with Eskenazi Health to waive fees for research patients to return for appointments in clinic. As it would be unethical to charge patients for research appointments, both facility and physician charges are waived. This helps patients defray costs for parking and travel, and significantly decreases the loss to follow-up.

This study represents a landmark multidisciplinary approach to prospective research at Eskenazi Health. The PI spent over a year recruiting and meeting with 30 IU clinical scientists from the disciplines of Orthopaedic Trauma, General Surgery, Anesthesiology, Physical Medicine & Rehab, and two IU PhD biostatistician. This protocol represents the consensus opinion of all of these faculty. The team consists of clinicians who prefer a conservative transfusion strategy, as well as those who prefer a more liberal transfusion strategy. The protocol was revised multiple times until all clinical scientists felt it was a safe and responsible approach to further study transfusion strategies in this young, healthy patient population.

The research team also consists of two full-time research coordinators, Valda Frizzell and Molly Moore, who have a cumulative experience of decades in participating in prospective studies such as this.

#### 12.0 References:

- 1. Leal-Noval, S.R., et al., *Transfusion of blood components and postoperative infection in patients undergoing cardiac surgery.* Chest, 2001. **119**(5): p. 1461-8.
- 2. Hebert, P.C., et al., A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med, 1999. **340**(6): p. 409-17.
- 3. Carson, J.L., et al., Risk of bacterial infection associated with allogeneic blood transfusion among patients undergoing hip fracture repair. Transfusion, 1999. **39**(7): p. 694-700.
- 4. Edna, T.H. and T. Bjerkeset, *Association between blood transfusion and infection in injured patients*. J Trauma, 1992. **33**(5): p. 659-61.

- 5. Hill, G.E., et al., *Allogeneic blood transfusion increases the risk of postoperative bacterial infection: a meta-analysis.* J Trauma, 2003. **54**(5): p. 908-14.
- 6. Vincent, J.L., et al., *Anemia and blood transfusion in critically ill patients*. JAMA, 2002. **288**(12): p. 1499-507.
- 7. Taylor, R.W., et al., *Impact of allogenic packed red blood cell transfusion on nosocomial infection rates in the critically ill patient.* Crit Care Med, 2002. **30**(10): p. 2249-54.
- 8. Leung, J.M., et al., *Electrocardiographic ST-segment changes during acute,* severe isovolemic hemodilution in humans. Anesthesiology, 2000. **93**(4): p. 1004-10.
- 9. Weiskopf, R.B., et al., *Human cardiovascular and metabolic response to acute, severe isovolemic anemia.* JAMA, 1998. **279**(3): p. 217-21.
- 10. Johnston, P., et al., *Is perioperative blood transfusion a risk factor for mortality or infection after hip fracture?* J Orthop Trauma, 2006. **20**(10): p. 675-9.

### **Appendix A: Screening Form**

| Sub | Subject ID: Date: | | |
|---|---|---|---|
| | Inclusion: (Must answer YES to all) | 1 | |
| 1. | Patients aged 18 to 50 years | ☐ Yes | □ No |
| 2. | Trauma patients admitted to participating hospital with any Orthopaedic injury who have been | □ Yes | □ No |
| | determined to be stable by the Trauma Service (General Surgery) and are no longer within the | | |
| | resuscitation phase of initial treatment. This is defined as a normal urine output (greater than 0.5 | | |
| | ml/kg/hr) and a systolic blood pressure greater than 90 mmHg for greater than 6 hours without | | |
| | fluid bolus or transfusion during that time | | |
| 3. | Hemoglobin less than 9 g/dL or expected drop below 9 g/dL with planned surgery | ☐ Yes | □ No |
| | Exclusion: (Must answer NO to all) | | |
| 1. | Women who are pregnant | ☐ Yes | □ No |
| 2. | Prisoner | ☐ Yes | □ No |
| 3. | Head injury(Glasgow Coma Scale less than 8 over 48 hours from presentation) | ☐ Yes | □ No |
| 4. | Known cardiac, renal (defined as having Serum Creatinine >1.2 at time of enrollment), liver, or | □ Yes | □ No |
| | pulmonary disease | | |
| 5. | Sickle cell anemia | ☐ Yes | □ No |
| 6. | History of cancer | ☐ Yes | □ No |
| 7. | Preexisting weakness, paresthesias, deformities, or other conditions which might affect functional outcome in the surgeon's opinion | ☐ Yes | □ No |
| 8. | Spinal cord injury | ☐ Yes | |
| 9. | Patients with burns expected to require operative treatment | ☐ Yes | |
| 10. | Unlikely to follow-up, as determined by the attending physician | ☐ Yes | |
| 11. | COVID positive | ☐ Yes | |
| 11. | COVID positive | res | |
| If v | ou answered yes to any of the exclusion items 1-11, the patient should be excluded. | | |
| 11 ) | ou answered <u>yes</u> to any of the exclusion fems 1-11, the patient should be excluded. | | |
| Pati | ent Enrollment Status: | | |
| | Included | | |
| | Excluded | | |
| | Refusal to consent (otherwise met inclusion/exclusion criteria) | | |
| | Inability to consent (otherwise met inclusion/exclusion criteria) | | |
| | Inability to consent (otherwise met inclusion/exclusion criteria) | | |

### **Appendix B: Patient Contact Form**

| Subject ID: | | Date:/ |
|---|---|---|
| Patient Name: | | DOB:/ |
| Address: | | City: |
| | Home Phone: ( ) - | Cell Phone: ( |
| Alternate Contact # 1 | - | |
| Name: | | Relationship to patient: |
| Address: | | City: |
| | Home Phone: () | Cell Phone: ( <u>)</u> - |
| Alternate Contact # 2 | | |
| Name: | | Relationship to patient: |
| Address: | | City: |
| Zip Code: | Home Phone: ( ) - | Cell Phone: ( <u>)</u> |
| | | · |

| Subject ID: | Date: / | / V | /isit Interval: 区 Pre-injury |
|-------------|---------|---------|--------------------------------|
| 345jeet 15: | Date | <b></b> | isic inicci van — i re injar y |

### Musculoskeletal Function Assessment

We would like you to answer the questions in this survey based on your condition <u>before</u> your injury.

Please answer "YES" or "NO" to each question by putting a check in the box  $\square$  next to the question. If the question was true for you <u>before</u> your injury, choose "YES". If the question was not true for you <u>before</u> your injury, choose "NO".

If you wish to comment on any of the questions, please use the space in the margins. Please answer all questions, even though some of the questions may not seem to apply to you.

| Subject ID: | Date: / | / V | /isit Interval: 区 Pre-injury |
|-------------|---------|---------|--------------------------------|
| 345jeet 15: | Date | <b></b> | isic inicci van — i re injar y |

| ACTIVITIES | USING TOUR | ARIVIS UR I | <u>.EG3</u> | | |
|---|---|---|---|---|---|
| This first set of questi carrying. <i>Before your</i> | | <u>r arms or legs</u> to do su | ch things as r | eaching | , walking, and |
| 1. Were you able to w | valk? | | | ☐ Yes | □ No |
| 2. Did you feel unstea | ady on your feet? | | | ☐ Yes | □ No |
| 3. Was it difficult for | you to reach up high? | | | ☐ Yes | □ No |
| 4. Did you straighten | or bend your arm(s) co | ompletely? | | ☐ Yes | □ No |
| 5. Did you straighten | or bend your leg(s) co | mpletely? | | ☐ Yes | □ No |
| 6. Did you pivot? | | | | ☐ Yes | □ No |
| 7. Did you climb up a | nd down ladders? | | | ☐ Yes | □ No |
| 8. Did you have to res | st often when walking? | <b>&gt;</b> | | ☐ Yes | □ No |
| 9. Did you avoid stairs | s? | | | ☐ Yes | □ No |
| 10. Did you stand for | long periods of time? | | | ☐ Yes | □ No |
| 11. Was it hard for you to get moving after you'd been sitting or lying down? | | | | | □ No |
| 12. Did you always walk with a limp? | | | | | □ No |
| 13. Did your leg some | etimes lock or give-way | /; | | ☐ Yes | □ No |
| 14. Did you have trou | ible getting in or out o | f a low chair? | | ☐ Yes | □ No |
| 15. Did you have trou | ible getting in or out o | f bed? | | ☐ Yes | □ No |
| 16. Did you kneel? | | | | ☐ Yes | □ No |
| 17. Did you pick up th | nings from the floor? | | | ☐ Yes | □ No |
| 18. Did you run at all? | | | | | □ No |
| 19. Did you have trouble getting in or out of a car? | | | | ☐ Yes | □ No |
| 20. Had you stopped using public transportation because of your physical | | | ohysical | ☐ Yes | . □ No |
| condition? Before your injury, ho (Please check one) | ow much were you bot | hered by problems usi | ng your arms | or legs? | ? |
| | □ 2 | □ 3 | □ 4 | | □ 5 |
| Not at A little Somewhat Quite Extremely all bothered bothered bothered bothered | | | | | Extremely |

Study #1402557771

| Subject ID: | | Date:/ | <u>/</u> | | Visit Interval | : ⊠ Pre-injury |
|---|---|---|---|---|---|---|
| <b>ACTIVITIES</b> | <u>USING YOUI</u> | R HANDS | | | | |
| The following question | ons are about activities | using your hands. <b>Bef</b> | ore your inju | ry | | ] |
| 1. Did you have diffic | ulty squeezing things? | | | ☐ Yes | □No | |
| 2. Could you make a | tight fist? | | | ☐ Yes | □ No | - |
| | u to put your hand in y | our pocket? | | ☐ Yes | □ No | |
| • | ulty turning knobs or l | • | ening | ☐ Yes | □ No | |
| 5. Did you have trouk | ole holding a book? | | | ☐ Yes | □ No | |
| 6. Did you have diffic | ulty writing or typing? | | | ☐ Yes | □ No | |
| 7. Did you have trouk | ole opening medicine b | oottles or jars? | | ☐ Yes | □ No | |
| Before your injury, ho | ow much were you bo | thered by problems us | ing your hand | ds? (Please | e check one) | _ |
| □ 1 | □ 2 | □ 3 | □ 4 | | □ 5 | |
| Not at all bothered | A little<br>bothered | Somewhat<br>bothered | Quite<br>bother | | Extremely bothered | |
| These questions are a | UND YOUR about activities around | l your home, including | such things a | as cooking | , cleaning, | ] |
| | with housework or ya | | | ☐ Yes | □No | |
| · | <u>,</u><br><u>h</u> housework or yard w | | | ☐ Yes | □ No | 1 |
| · | you to do household c | • | ok so <u>much</u> | ☐ Yes | □ No | |
| 4. Did you mop or sw | reep or vacuum? | | | ☐ Yes | □ No | |
| 5. Was scrubbing a pan or dish difficult? | | | | | □ No | |
| 6. Did you need some | eone to cook for you? | | | ☐ Yes | □ No | |
| 7. Did it take you a <u>lo</u> | ng time to do househo | old chores? | | ☐ Yes | □ No | |
| | you to shop for grocer<br>loing car, house, or ma | | ause of | ☐ Yes | □ No | - |

Study #1402557771 v. 07/31/2020

your physical condition?

☐ Yes

☐ No

| Subject ID: | | Date:/ | / | | Visit Interval: | ⊠ Pre-injury |
|---|---|---|---|---|---|---|
| Before your injury, ho | ow much were you bot | thered by problems do | ing work arou | ınd your | home? (Please ch | eck one) |
| ☐ 1 Not at all bothered | ☐ 2 A little bothered | ☐ 3 Somewhat bothered | ☐ 4<br>Quite<br>bothere | | ☐ 5 Extremely bothered | |
| SELF CARE | | | | | | |
| The following question | ons are about <u>taking ca</u> | are of yourself. <b>Before</b> | your injury | | | |
| 1. Did you wear thing | s that were easier to g | get into? | | ☐ Yes | □ No | |
| 2. Did you sometimes | s_need help from other | rs to get dressed? | | ☐ Yes | □ No | |
| 3. Did you struggle w | ith buttons, snaps, hoo | oks, zippers? | | ☐ Yes | □ No | |
| 4. Did you have troub | ole pulling clothes on o | ver your head? | | ☐ Yes | □ No | |
| 5. Was it difficult for | you to put on shoes, s | ocks, or stockings? | | ☐ Yes | □ No | |
| 6. Was it a chore for | you to dress because i | t took so long? | | ☐ Yes | □ No | |
| 7. Was it difficult to b | orush your teeth? | | | ☐ Yes | □ No | |
| 8. Did you have a diff | icult time cutting your | fingernails? | | ☐ Yes | □ No | |
| 9. Did you need help | keeping yourself clear | after going to the bat | hroom? | ☐ Yes | □ No | |
| 10. Was it difficult for | r you to get on or off t | he toilet? | | ☐ Yes | □ No | |
| 11. Was it hard for yo | ou to get in or out of th | ne bathtub or shower? | | ☐ Yes | □ No | |
| 12. Did you sit while | showering? | | | ☐ Yes | □ No | |
| 13. Did you need help | o washing yourself? | | | ☐ Yes | □ No | |
| 14. Did you need help eating? | | | | | □ No | |
| 15. Was it hard for you to cut food? | | | | | □ No | |
| 16. Were you stuck at home because of your physical condition? | | | | | □ No | |
| 17. Had you stopped going out by yourself? | | | | | □ No | |
| 18. Had you stopped driving because of your physical condition? | | | | ☐ Yes | □ No | |
| Before your injury, ho | ow much were you bot | thered by problems ca | ring for yours | elf? <i>(Ple</i> | ase check one) | 1 |
| ☐ 1 | ☐ 2 | ☐ 3 | ☐ 4 | | ☐ 5 | |
| Not at A little Somewhat Qui | | | | | Extremely | |

| Subject ID: | | Date:/ | <i>J</i> | | Visit Interval: | ⊠ Pre-injury |
|---|---|---|---|---|---|---|
| SLEEP AND | <u>REST</u> | | | | | |
| These questions are a your injury | about changes or prob | lems you may have ex | perienced wit | th <u>sleep a</u> | and rest. <b>Before</b> | |
| 1. Were you tired all | of the time? | | | ☐ Yes | □No | |
| 2. Did you have trouk | ole falling asleep at nig | ht? | | ☐ Yes | □ No | |
| 3. Did you have diffic | ulty sleeping the whole | e night? | | ☐ Yes | □ No | |
| 4. Was it hard for you | u to get comfortable to | sleep? | | ☐ Yes | □ No | |
| 5. Did you wake up s | ooner than you would | like? | | ☐ Yes | □ No | |
| 6. Did you have distu | rbing dreams? | | | ☐ Yes | □ No | |
| Before you injury ho | w much were you botl | nered by problems wit | h sleen and r | est? (Plei | ase check one) | |
| | | □ 3 | | | □ 5 | |
| Not at | A little | Somewhat | Quite | | Extremely | |
| all bothered | bothered | bothered | bother | ed | bothered | |
| LEISURE an | d RECREATION | ONAL ACTIV | <u>ITIES</u> | | | |
| leisure time or recrea | ons are about changes<br>ational activities. These<br>or volunteering. <b>Befor</b> e | activities may include | | | | |
| | fitness worse because | | sical | ☐ Yes | □ No | |
| 2. Did you do <u>less</u> of your usual physical recreational activities because of your health or physical condition? | | | | | □ No | |
| 3. Had you stopped o | loing <u>all</u> of your usual <sub>l</sub> | ohysical recreational a | ctivities? | ☐ Yes | □ No | |
| 4. Were you doing fewer leisure activities (such as hobbies, crafts, gardening, card playing, going out with friends) because of your health or physical | | | | | □ No | |
| condition? | | | | | | |
| Before your injury, ho | ow much were you bo | thered by problems do | ing leisure ar | nd recrea | tional activities? (P | lease check |
| □ 1 | □ 2 | □ 3 | □ 4 | | □ 5 | |
| Not at all bothered | A little<br>bothered | Somewhat<br>bothered | Quite<br>bother | | Extremely bothered | |

| Subject ID: | | Date:/ | / | | Visit Interva | ıl: 🗵 Pre-injur |
|---|---|---|---|---|---|---|
| <b>RELATIONS</b> | HIPS: FAMIL | Y and FRIEN | <u>DS</u> | | | |
| | | 6 6 | | | | $\neg$ |
| life. <i>Before your inju</i> | | os with family, friends, | and other in | portant | t people in your | |
| 1. Was there a strain | in your relationships v | vith either your friends | or family? | ☐ Yes | s □ No | |
| | st didn't want to be ar | | | ☐ Yes | S □ No | |
| 3. Was it hard for you things? | ı to get either your fan | nily or friends to help y | ou do | ☐ Yes | s □ No | |
| 4. Were you lonely? | | | | ☐ Yes | s □ No | |
| - | • | mily had shied away fr | | ☐ Yes | S □ No | |
| • | rritable towards those<br>swers, criticize easily) | around you (for exam | ple, snap at | ☐ Yes | S □ No | |
| 7. Did you miss being | with either your frien | ds or family? | | ☐ Yes | s □ No | |
| 8. Did you feel like be | eing less intimate beca | use of your physical co | ndition? | ☐ Yes | S □ No | |
| 9. Had your sexual lif | e changed because of | your physical condition | 1? | ☐ Yes | S □ No | |
| 10. Did you enjoy sex | less because of your p | physical condition? | | ☐ Yes | S □ No | |
| Before your injury, ho<br>people in your life? (I | • | thered by problems yo | u had with yo | our frien | ids, family, and ot | ner important |
| □ 1 | □ 2 | □ 3 | □ 4 | | □ 5 | |
| Not at all bothered | A little<br>bothered | Somewhat<br>bothered | Quite<br>bother | | Extremely bothered | |
| an bothered | bothered | bothered | botner | eu | bothered | _ |
| <b>THINKING</b> | | | | | | |
| These questions are a | about <u>thinking, concer</u> | trating, or rememberi | ng. <i>Before yo</i> | ur injur | y | |
| 1. Did it take you a lo | ng time to figure thing | s out? | | ☐ Yes | S □ No | |
| 2. Did you have problems with concentration? | | | | | S □ No | |
| 3. Were you confused and scattered? | | | | | S □ No | |
| 4. Were you forgetful? | | | | | S □ No | |
| Before your injury, ho | ow much were you bo | thered by problems wi | th thinking, c | oncentr | ating, and remem | bering? <i>(Please</i> |
| □ 1 | □ 2 | □ 3 | □ 4 | | □ 5 | |
| Not at all bothered | A little<br>bothered | Somewhat<br>bothered | Quite<br>bother | | Extremely bothered | |

| Subject ID: | | Date:/ | _/ | | Visit Interval: | ☑ Pre-injury |
|---|---|---|---|---|---|---|
| LIFE CHANG | SES and FEEL | <u>.INGS</u> | | | | |
| The following questic | ons are about the day | • • | | u may hav | ve been | |
| | s use your physical cor | | | ☐ Yes | □ No | |
| 2. Did you have to co | ncentrate when using | your hands, arms, le | gs, or feet? | ☐ Yes | □ No | |
| 3. Did you avoid using | g your hands, arms, le | gs, or feet? | | ☐ Yes | □ No | |
| 4. Did you protect yo | ur hands, arms, legs, c | or feet? | | ☐ Yes | □ No | |
| 5. Did you accept you | physical condition? | | | ☐ Yes | □ No | |
| 6. Did you feel your li condition? | fe had changed becau | se of your health or p | ohysical | ☐ Yes | □ No | |
| 7. Did you feel your p | hysical condition was | getting worse over ti | me? | ☐ Yes | □ No | |
| 8. If you did too much | n in one day, did it affe | ect what you did the i | next day? | ☐ Yes | □ No | |
| 9. Did you feel disable | ed, even though you n | nay have looked fine | to others? | ☐ Yes | □ No | |
| 10. Did you feel usele | ess? | | | ☐ Yes | □ No | |
| 11. Did you feel unat | tractive? | | | ☐ Yes | □ No | |
| 12. Did your physical | condition make you fe | eel less capable? | | ☐ Yes | □ No | |
| 13. Did you feel sorry for yourself? | | | | | □ No | |
| 14. Did you feel like you complained a lot? | | | | | □ No | |
| 15. Did you have to ask for help a lot? | | | | ☐ Yes | □ No | |
| 16. Did you feel angry or frustrated about your health or any physical condition? | | | ☐ Yes | □ No | | |
| Before your injury, howere experiencing in | ow much were you bo<br>your life? | thered by the day to | day adjustmer | nts you we | ere making and the | e feelings you |
| □ 1 | □ 2 | □ 3 | | 1 | □ 5 | |

Study #1402557771 v. 07/31/2020

Somewhat

bothered

Quite

bothered

Extremely bothered

A little

bothered

Not at

all bothered

| Subject ID: | | Date:/ | / | | Visit Interval: | 区 Pre-injur |
|---|---|---|---|---|---|---|
| WORK ACT | <u>IVITIES</u> | | | | | |
| Were you working be | efore you injury? | | | | | |
| □ NoWe | ere you unable to work | because of your healt | h or physical | conditio | n? | |
| | □No | | | | | |
| | □Yes | | | | | |
| □Yes (plo | ease answer the quest | ions below) | | | | |
| | | | | | | ٦ |
| Please answer these your injury | questions as they desc | ribe your experiences | at work befo | re your i | injury. <i>Before</i> | |
| 1. Were you making | changes in your joh? | | | ☐ Yes | s □ No | |
| • | ult for you to do your jo | ob because of your hea | alth or | ☐ Yes | | |
| 3. Were you slow at your job because of your health or physical condition? | | | | | | |
| 4. Did you take more breaks because of your health or physical condition? | | | | | | |
| Before your injury, he | ow much were you bo | thered by problems wi | th work activ | vities, be | cause of your physi | cal condition? |
| □ 1 | □ 2 | □ 3 | | 1 | □ 5 | |
| Not at | A little | Somewhat<br>bothered | Quite<br>bother | | Extremely bothered | |

| Subject ID: | Date:/ | Visit Interval: ☐ 6month ☐ 1 year |
|-------------|--------|-----------------------------------|
|-------------|--------|-----------------------------------|

### Musculoskeletal Function Assessment

We are interested in finding out how you are managing with your injury or arthritis this week.

Please answer "YES" or "NO" to each question by putting a check in the box □ next to the question. If the question was true for you and is related to your injury or arthritis, choose "YES". If the question was not true for you and is not related to your injury or arthritis, choose "NO".

If you wish to comment on any of the questions, please use the space in the margins. Please answer all questions, even though some of the questions may not apply to your injury or arthritis.

### FA)

| Subject ID: | | Visit | Interval: 6month | □ 1 ye |
|---|---|---|---|---|
| <b>ACTIVITIES USING</b> | YOUR ARMS OR LEGS | | | |
| | changes or problems you may have <u>using yo</u><br>arrying. <i>This week, because of your injury or</i> | | | |
| 1. Are you able to walk? | | ☐ Yes | □ No | |
| 2. Do you feel unsteady on your fe | eet? | ☐ Yes | □ No | |
| 3. Is it difficult for you to reach up | high? | ☐ Yes | □ No | |
| 4. Do you straighten or bend your | arm(s) completely? | ☐ Yes | □ No | |
| 5. Do you straighten or bend your | leg(s) completely? | ☐ Yes | □ No | |
| 6. Do you pivot? | | ☐ Yes | □ No | |
| 7. Do you climb up and down ladd | ers? | ☐ Yes | □ No | |
| 8. Do you have to rest often when | walking? | ☐ Yes | □ No | |
| 9. Do you avoid stairs? | | ☐ Yes | □ No | |
| 10. Do you stand for long periods | of time? | ☐ Yes | □ No | |
| 11. Was it hard for you to get mov | ring after you'd been sitting or lying down? | ☐ Yes | □ No | |
| 12. Do you always walk with a lim | 0? | ☐ Yes | □ No | |
| 13. Do your legs sometimes lock o | r give-way? | ☐ Yes | □ No | |
| 14. Do you have trouble getting in | or out of a low chair? | ☐ Yes | □ No | |
| 15. Do you have trouble getting in | or out of bed? | ☐ Yes | □ No | |
| 16. Do you kneel? | | ☐ Yes | □ No | |
| 17. Do you pick up things from the | e floor? | ☐ Yes | □ No | |
| 18. Do you run at all? | | ☐ Yes | □ No | |
| 19. Do you have trouble getting in | or out of a car? | ☐ Yes | □ No | |
| 20. Had you stopped using public condition? | transportation because of your physical | ☐ Yes | □ No | |

(Please check one)

| □ 1 | □ 2 | □ 3 | □ 4 | □ 5 |
|--------------|----------|----------|----------|-----------|
| Not at | A little | Somewhat | Quite | Extremely |
| all bothered | bothered | bothered | bothered | bothered |

| Subject ID: | | Date:/ | | ٧ | 'isit Interval: ☐ 6m | onth 🗆 1 year |
|---|---|---|---|---|---|---|
| ACTIVITIES USING YOUR HANDS | | | | | | |
| | | | | | | ı |
| arthritis | ons are about activities | s <u>using your</u> nands. <i>T</i> i | піѕ wеек, реса | use of y | our injury or | 1 |
| 1. Do you have difficu | ulty squeezing things? | | | ☐ Yes | □ No | 1 |
| 2. Do you have difficu | ulty making a tight fist? | ? | | ☐ Yes | □ No | 1 |
| 3. Is it hard for you to | put your hand in you | r pocket? | | ☐ Yes | □ No | ı |
| 4. Do you have difficution folling down car wind | ulty turning knobs or le<br>dows)? | evers (for example, o | pening doors, | ☐ Yes | □ No | 1 |
| 5. Do you have troub | | | | ☐ Yes | □ No | 1 |
| 6. Do you have difficu | ulty writing or typing? | | | ☐ Yes | □ No | 1 |
| 7. Do you have troub | le opening medicine b | ottles or jars? | | ☐ Yes | s □ No | ı |
| How much are you be | othered by problems y | ou are <b>now</b> having u | sing your hand | ls? (Plea | se check one) | |
| | | | | | □ 5 | |
| Not at | A little | Somewhat | Quite | | Extremely | |
| all bothered | bothered | bothered | bother | ed | bothered | |
| WORK ARO | UND YOUR | <u>HOME</u> | | | | |
| · | about <u>activities around</u><br>airs. <b>This week, becaus</b> | • | - | as cookir | ng, cleaning, | ı |
| | with housework or yar | | | ☐ Yes | □ No | 1 |
| | n housework or yard w | | | ☐ Yes | □ No | 1 |
| · | old chores but find tha | | :? | ☐ Yes | □ No | 1 |
| 4. Do you mop or swe | | | - | ☐ Yes | □ No | 1 |
| 5. Is scrubbing a pan | or dish difficult? | | | ☐ Yes | □ No | 1 |
| 6. Do you need some | one to cook for you? | | | ☐ Yes | □ No | 1 |
| 7. Does it take you <u>lo</u> | nger to do household | chores? | | ☐ Yes | s □ No | 1 |
| 8. Is it difficult for you to shop for groceries or other thing? | | | | | | |
| 9. Have you stopped doing car, house, or maintenance repairs because of your injury or arthritis? | | | | | | |
| How much are vou be | othered by problems y | ou are <b>now</b> having d | oing work aro | und vour | home? (Please che | ck one) |
| □ 1 | □ 2 | □ 3 | | • | □ 5 | , |
| Not at | A little | Somewhat | Quite | | | |
| all bothered | bothered | bothered | bother | | bothered | |

Study #1402557771 v. 07/31/2020

| Subject ID: | | Date:/ | J | Vi | sit Interval: 🗆 6m | onth 🗆 1 year |
|---|---|---|---|---|---|---|
| SELF CARE | <u>ACTIVITIES</u> | | | | | |
| The following question. | ons are about taking ca | are of yourself. <i>This w</i> | eek, because | of your ii | njury or arthritis . | |
| 1. Do you wear thing | s that are easier to get | into? | | ☐ Yes | □ No | |
| 2. Do you <u>sometimes</u> | _need help from other | s to get dressed? | | ☐ Yes | □ No | |
| 3. Do you struggle wi | th buttons, snaps, hoo | ks, zippers? | | ☐ Yes | □ No | |
| 4. Do you have troub | le pulling clothes on o | ver your head? | | ☐ Yes | □ No | |
| 5. Is it difficult for you | u to put on shoes, sock | ks, or stockings? | | ☐ Yes | □ No | |
| 6. Is it a chore for you | u to dress because it to | ook so long? | | ☐ Yes | □ No | |
| 7. Is it difficult to bru | sh your teeth? | | | ☐ Yes | □ No | |
| 8. Do you have a diffi | cult time cutting your | fingernails? | | ☐ Yes | □ No | |
| 9. Do you need help l | keeping yourself clean | after going to the bat | throom? | ☐ Yes | □ No | |
| 10. Is it difficult for yo | ou to get on or off the | toilet? | | ☐ Yes | □ No | |
| 11. Is it hard for you | to get in or out of the I | bathtub or shower? | | ☐ Yes | □ No | |
| 12. Do you sit while s | howering? | | | ☐ Yes | □ No | |
| 13. Do you need help | washing yourself? | | | ☐ Yes | □ No | |
| 14. Do you need help | eating? | | | ☐ Yes | □ No | |
| 15. Is it hard for you | to cut food? | | | ☐ Yes | □ No | |
| 16. Are you stuck at h | nome? | | | ☐ Yes | □ No | |
| 17. Have you stopped | d going out by yourself | ? | | ☐ Yes | □ No | |
| 18. Have you stopped driving because of your physical condition? | | | | | □ No | |
| This week, because of your injury or arthritis, how much were you bothered by problems caring for yourself? (Please check one) | | | | | | |
| □ 1 | □ 2 | □ 3 | □ 4 | | □ 5 | |
| Not at<br>all bothered | A little<br>bothered | Somewhat<br>bothered | Quite<br>bother | | Extremely bothered | |

| Subject ID: | <del></del> | Date:/ | / | V | isit Interval: 🗆 6m | onth $\square$ 1 year |
|---|---|---|---|---|---|---|
| <b>SLEEP AND</b> | REST | | | | | |
| • | about changes or prob<br>ur injury or arthritis | | riencing with | sleep ar | nd rest. <i>This</i> | |
| 1. Are you tired all of | the time? | | | ☐ Yes | □No | |
| 2. Do you have troub | le falling asleep at nigh | nt? | | ☐ Yes | □ No | |
| 3. Do you have difficu | ulty sleeping the whole | e night? | | ☐ Yes | □ No | |
| 4. Is it hard for you to | get comfortable to sl | eep? | | ☐ Yes | □ No | |
| 5. Do you wake up so | oner than you would l | ike? | | ☐ Yes | □ No | |
| 6. Do you have distur | bing dreams? | | | ☐ Yes | □ No | |
| How much are you bo | othered by problems y | ou are <u>now</u> having wit | :h sleep and r | est? (Ple | ease check one) | |
| □ 1 | □ 2 | □ 3 | □ 4 | | □ 5 | |
| Not at all bothered | A little<br>bothered | Somewhat<br>bothered | Quite<br>bother | | Extremely bothered | |
| We would also like to activities. These activ | o know about changes rities may include such the cek, because of your in | or problems you are h<br>things as hobbies, spo | aving with <u>lei</u> | | | |
| | ness worse because of | | I | ☐ Yes | □ No | |
| | our usual physical recoal condition? | reational activities bec | ause of | ☐ Yes | □ No | |
| | doing <u>all</u> of your usual | | | ☐ Yes | □ No | |
| 4. Are you doing fewer leisure activities (such as hobbies, crafts, gardening, card playing, going out with friends) because of your health or physical condition? | | | | | | |
| How much are you bo | othered by problems y | ou are <b>now</b> having wit | :h leisure and | recreati | ional activities? (Ple | ease check one |
| □ 1 | □ 2 | ☐ 3 | □ 4 | | □ 5 | - <b>-</b> / |
| Not at<br>all bothered | A little<br>bothered | Somewhat<br>bothered | Quite<br>bother | | Extremely bothered | |

| Subject ID: | ····· | Date:/ | / | V | isit In | terval: 🗆 6m | onth 🗆 1 year |
|---|---|---|---|---|---|---|---|
| <b>RELATIONS</b> | HIPS: FAMIL | Y and FRIEN | <u>DS</u> | | | | |
| Those questions are | about your <u>relationshi</u> j | as with family friends | and other im | nortant | noon | lo in vour | |
| | use of your injury or a | | and other in | iportani | peop | <u>le</u> ili youi | |
| 1. Is there a strain in | your relationships with | n either your friends o | family? | ☐ Yes | | □ No | |
| 2. Do you feel you jus | st don't want to be arc | ound anybody? | | ☐ Yes | | □ No | |
| 3. Is it hard for you to | get either your family | or friends to help you | ı do things? | ☐ Yes | | □ No | |
| 4. Are you lonely? | | | | ☐ Yes | | □ No | |
| | ther your friends or fa | | | ☐ Yes | | □ No | |
| · | ritable towards those assily) | | ole, snap at | ☐ Yes | | □ No | |
| 7. Do you miss being | with either your friend | ds or family? | | ☐ Yes | | □ No | |
| 8. Do you feel like be | ing less intimate? | | | ☐ Yes | | □ No | |
| 9. Has your sexual life | e changed? | | | ☐ Yes | | □ No | |
| 10. Do you enjoy sex | less? | | | ☐ Yes | | □ No | |
| How much are you be your life? (Please che | othered by problems y | ou are <u>now</u> having wit | h your friend | s, family | , and | other importa | int people in |
| □ 1 | □ 2 | □ 3 | □ 4 | | | □ 5 | |
| Not at | A little | Somewhat | Quite | | | Extremely bothered | |
| all bothered | bothered | bothered | bother | eu | L. | otherea | |
| <b>THINKING</b> | | | | | | | |
| These questions are a or arthritis | about thinking, concen | trating, or rememberi | ng. <b>This week</b> | k, becau | se of y | our injury | |
| 1. Does it take you a | long time to figure thir | ngs out? | | ☐ Yes | | □ No | |
| 2. Do you have probl | ems with concentratio | ☐ Yes | | □ No | | | |
| 3. Are you confused and scattered? | | | | | | | |
| 4. Are you more forgetful? ☐ Yes ☐ No | | | | | | | |
| How much are you be | othered by problems y | ou are <u>now</u> having thi | nking, concer | ntrating, | and re | emembering? | (Please check |
| □ 1 | □ 2 | □ 3 | □ 4 | | | □ 5 | |
| Not at all bothered | A little<br>bothered | Somewhat<br>bothered | Quite<br>bother | | | xtremely<br>othered | |

Study #1402557771

| Subject ID: | | Date:/_ | | | V | isit In | terval: 🗆 6m | onth □ 1 year |
|---|---|---|---|---|---|---|---|---|
| LIFE CHANG | SES and FEEL | <u>INGS</u> | | | | | | |
| • | These questions are about the <u>day to day adjustments</u> you may be making because of your injury or arthritis and <u>feelings</u> you may be having about your experiences. <i>This week, because of your injury or arthritis</i> | | | | | | | |
| 1. Do you sometimes things? | use your physical cond | dition as an excuse | not to do | | ☐ Yes | | □ No | |
| 2. Do you have to cor joints? | ncentrate when using y | our injured limb o | r arthritic | | ☐ Yes | | □ No | |
| 3. Do you avoid using | your injured limb or a | rthritic joints? | | | ☐ Yes | | □ No | |
| 4. Do you protect you | ır injured limb or arthr | itic joints? | | | ☐ Yes | | □ No | |
| 5. Do you think every | thing will work out in t | the long run? | | | ☐ Yes | | □ No | |
| 6. Do you accept you | r current situation? | | | | □ Yes | | □ No | |
| 7. Do you feel everytl | ning is back to normal? | ) | | | □ Yes | | □ No | |
| 8. Do you feel your lif | e has changed quite a | bit? | | | □ Yes | | □ No | |
| 9. Are you getting wo | rse? | | | | ☐ Yes | | □ No | |
| 10. If you do too muc | h in one day, does it a | ffect what you do t | he next da | ay? | ☐ Yes | | □ No | |
| 11. Do you feel disab | led, even though you r | nay look fine to oth | ners? | | ☐ Yes | | □ No | |
| 12. Do you feel usele | ss? | | | | ☐ Yes | | □ No | |
| 13. Do you feel unatt | ractive? | | | | ☐ Yes | | □ No | |
| 14. Does your injury o | or arthritis make you fe | eel less capable? | | | ☐ Yes | | □ No | |
| 15. Do you feel sorry | for yourself? | | | | ☐ Yes | | □ No | |
| 16. Do you feel like you complained a lot? | | | | | ☐ Yes | | □ No | |
| 17. Do you have to ask for help a lot? | | | | | ☐ Yes | | □ No | |
| 18. Do you feel angry or frustrated that you have this injury or arthritis? | | | | | ☐ Yes | | □ No | |
| • | How much are you bothered by the day to day adjustments you are making in your life and the feelings you are now experiencing, because of your injury or arthritis? (Please check one) | | | | | | ou are <u>now</u> | |
| ☐ 1<br>Not at | □ 2<br>A little | ☐ 3<br>Somewhat | | ☐ 4<br>Quite | | E | ☐ 5<br>ctremely | |

bothered

bothered

all bothered

bothered

bothered

| Subject ID: | | Date:/ | / | Visit Interval: $\square$ 6month $\square$ 1 year | | |
|---|---|---|---|---|---|---|
| <b>WORK ACT</b> | IVITIES | | | | | |
| Are you working now | <u>'?</u> | | | | | |
| ☐ NoAre | you unable to work b | ecause of your injury o | or arthritis? | | | |
| ☐No (Please skip to the next section) | | | | | | |
| | □Yes (Please skip t | to the next section) | | | | |
| □Yes (Ple | ease answer the quest | ions below) | | | | |
| Please answer these injury or arthritis | questions as they desc | ribe your experiences | at work. <i>This</i> u | week, be | cause of your | |
| 1. Are you making ch | anges in your job? | | | □ Yes | □ No | |
| 2. Is it more difficult | for you to do your job | now? | | ☐ Yes | □ No | |
| 3. Are you slower at y | your job? | | | ☐ Yes | □ No | |
| 4. Do you take more | breaks? | | | □ Yes | □ No | |
| How much are you be (Please check one) | othered by problems y | ou are <u>now</u> having wit | h work activiti | ies, beca | use of your injury | or arthritis? |
| □ 1 | □ 2 | □ 3 | □ 4 | | □ 5 | |
| Not at | A little | Somewhat | Quite | 4 | Extremely | |

Study #1402557771 v. 07/31/2020

| Subjec | ct ID: Visit Interval: $\square$ 6month $\square$ 1 year |
|---|---|
| | have completed this survey before, please answer the following three questions. If you ompleting this survey for the first time, please skip them. |
| 1. | Have you had any injuries or other important changes in your health since you completed the <u>last</u> survey? ☐ No |
| | ☐ Yes If yes, please list whatever injuries or health changes you have had: |
| 2. | Have you had any surgeries or hospitalizations since you completed the <u>last</u> survey? ☐ No |
| | ☐ Yes If yes, please list whatever injuries or health changes you have had: |
| 3. | How is your injury or arthritis <u>now,</u> compared to when you completed the <u>last</u> survey? <i>(Check one)</i> Much worse |
| | Slightly worse□ |
| | About the same |
| | Slightly better□ |
| | Much better |

### Appendix E: 2 Minute Walk Test

| Data: / | / | aniatawa T | | | 0.07. |
|---|---|---|---|---|---|
| | | | | | 02 %: |
| | e Used: | | | | |
| | | ik: BP: _ | / | O <sub>2</sub> | Vitals after test: HR: _ |
| BP:/Pt unable to comp | | | | | |
| | ing OR/on bed rest | | | | |
| ∐ Physic | cal inability to complete | due clinical indication | on such as | pain/decre | ase in vitals. |
| Completed by: _ | | | | | |
| | | _ | | | |
| Date:/ | / | Assistance Level: _ | | | 02 %: |
| Assistive Device | e Used: | | Distai | nce ambula | ted in 2 minutes: |
| | | | | | Vitals after test: HR: _ |
| BP:/ | O <sub>2</sub> | | | | |
| Pt unable to comp | plete test due to: | | | | |
| ☐ Pend | ing OR/on bed rest | | | | |
| ☐ Physic | cal inability to complete | due clinical indication | on such as | pain/decre | ase in vitals. |
| Completed by: | | | | | |
| completed by: _ | | | | | |
| | , | <u>-</u> | | | |
| Date:/ | | Assistance Level: _ | | | |
| | e Used: | | | | |
| | | IR: BP: _ | / | O <sub>2</sub> | Vitals after test: HR: _ |
| BP:/ | <del></del> | | | | |
| Pt unable to comp | | | | | |
| □ Pend | ing OR/on bed rest | | | | |
| ☐ Physic | cal inability to complete | due clinical indication | on such as | pain/decre | ase in vitals. |

### Appendix E: 2 Minute Walk Test

| Subject ID: |
|---------------|
| Completed by: |

### Appendix F: Adverse Event

| oject II | | $ \Box \ 6 \ \text{months} \ \Box \ 9 \\ \text{months} \ \Box \ 1 \\ $ | Report Date:// |
|---|---|---|---|
| | eate of event:// | | year |
| | Osteomyelitis | Urinary tract infection | □ Pneumonia |
| | Renal insufficiency | Cardiac ischemia | ☐ Myocardial infarction |
| | Deep venous thrombosis □ | Reoperation | ☐ Re-hospitalization (//) |
| | Infection | | |
| | ☐ Superficial (cellulitis treate | ed with oral antibiotics) | |
| | ☐ Deep (requires IV antibiot | ics or surgical debridement) | |
| | Other: | | |
| <b>P</b> 1 | lease list any details of event | | |
| _ | lease list any details of event. | | |
| E | vent related to treatment? | | |
| | ☐ Related ☐ Probabl | y Related □Possibly Related | □ Not Related |
| C | lassification of AE: | | |
| | □ Expected | | |
| | ☐ Unexpected | | |
| | □Serious (check below) | | |
| | □Requires/prolon | gs inpatient hospitalization | |
| | ☐ Immediately lif | e-threatening | |
| | □Permanently dis | abled | |
| | $\Box$ Fatal | | |
| O | outcome: | | |
| | ☐ Resolveddate resol | ved/ | |
| | ☐ Resolved with impairm | nentdate resolved/ | / |
| | Degree of impair | ment: □ Mild □ Moderate □Seve | ere |
| | $\Box$ Ongoing | | |

### **Appendix G: Protocol Deviation**

| ubject ID: | Report Date: | / | / |
|----------------------------------------|--------------|---|---|
| 1. Date of deviation:/ | | | |
| 2. Please describe protocol deviation: | | | _ |

### Appendix H: Escape Criteria

| ıbject ID: | | | Report Date: | / | |
|---|---|---|---|---|---|
| 1. Transfusion T | `ime:: | | | | |
| | was transfused: | | | | |
| ☐ Patient has | any of the following s | ymptoms at rest: chest pai | n, shortness of breath, dizzi | ness | |
| ☐ Patient has | a mean arterial pressur | re less than 50 mmHg that | is not responsive to fluid re | esuscitation | n |
| ☐ At any time | the patient's heart rat | e increases by more than 3 | 30% above baseline while u | nder anestl | hesia |
| ☐ The patient rehydration with | | o less than 0.5 mL/kg/hou | r and remains decreased des | spite adequ | ıate |
| | serum cardiac marker | | ollowing: EKG changes such<br>an 6, lactate greater than 2.5 | | |
| | in systolic blood press<br>luid resuscitation | ure by 10% or more with | exercise (physical therapy) | that does r | ıot |
| ☐ Uncontrolle | ed source of hemorrhage | ge | | | |
| ☐ Asympton | natic- Hgb dropped b | elow randomization thr | reshold | | |
| 3. Lowest Hgb pr | ior to transfusion: | g/dL | | | |

### Appendix H: Escape Criteria

| Sub | ect ID: | Report Date: / / |
|-----|-----------|------------------|
| Jub | nject iD. | Report Date. |

### **Appendix I: Length of Stay**

| Subject ID: | | Report Date:// |
|--------------------------------|------|----------------|
| Date of hospital admission: | | |
| 2. Date of hospital discharge: | / | |
| 3 Length of hospital stay: | days | |

## Appendix J: American Academy of Orthopaedic Surgeons Abstract February 2011 San Diego, CA (Podium Presentation)

Does Anemia or Transfusion Increase the Risk of Complications in Orthopaedic Trauma Patients?

Introduction: Transfusion of young, healthy, asymptomatic Orthopaedic trauma patients is routine at many institutions due to concerns for anemia. The purpose of this study is to assess whether anemia, with or without allogeneic blood transfusion, contributes to an increased complication rate in healthy orthopaedic trauma patients and whether the transfusion itself might be an independent risk factor for a complication.

Methods: A retrospective review of 104 patients treated at a level-one trauma center from September 2006-February 2009 was conducted. Inclusion criteria were patients 18-50 years of age, a hemoglobin concentration of 9.0 g per deciliter (g/dL) or less at any time during their admission. Head injured patients or patients with history or pulmonary or cardiac conditions were excluded. The patients were initially divided into two cohorts by their lowest hemoglobin level prior to first transfusion of < 7.0 (g/dl) and >7.0 (g/dl); this was followed by further division depending on whether the patients were transfused. Logistic regression analysis was performed.

Results: There was no increased risk for complication related to anemia itself (p=0.3). However, there was a significant risk for complication related to transfusion (p<0.01); furthermore, there was a dose-dependent effect with complication risk increasing with each unit transfused (p=0.02). Other factors such as age, injury severity score (ISS), and gender were considered and when adjusted did not change these results.

Conclusion: In young, healthy Orthopaedic trauma patients anemia does not appear to act as an independent risk factor for complications; however, allogeneic blood transfusion does appear to be a significant independent risk factor for complication and has a dose-dependent effect.

#### Appendix K: American Journal of Orthopaedics, 2015

Does Anemia or Transfusion Increase the Risk of Complications in Orthopaedic Trauma Patients? Mullis BH, Fisk E, Weaver D, Zhao Q, Daggy J Indiana University School of Medicine Department of Orthopaedics

**Introduction:** Transfusion of young, healthy, asymptomatic Orthopaedic trauma patients is routine at many institutions due to concerns for anemia. The purpose of this study was to assess whether anemia, with or without allogeneic blood transfusion, contributed to an increased complication rate in healthy Orthopaedic trauma patients and whether the transfusion itself might be an independent risk factor for a complication.

**Methods**: A retrospective review of 104 patients treated at a level 1 trauma center by a single surgeon from September 2006- February 2009 was conducted. Inclusion criteria were patients 18-50 years of age and a hemoglobin concentration of 9.0 g per deciliter (g/dL) or less at any time during their admission. Patients with head injury, pregnancy, or patients with a pre-existing history of pulmonary, cardiac, or renal conditions were excluded. The patients were initially divided into two cohorts by their lowest hemoglobin level prior to first transfusion of < 7.0 (g/dl) and > 7.0 (g/dl); this was followed by further division depending on whether the patients were transfused. Logistic regression analysis was performed. Patients' charts were reviewed for complications extending through a one-year period after initial discharge from the inpatient service. Patients who had not received follow-up treatment through a known outpatient clinic were contacted by telephone to ascertain outcome. Overall, 5 out of 104 patients were lost at one-year follow-up. Among other variables, postoperative complications were recorded as our primary outcome. Superficial wound infection was defined as cellulitis within one year requiring oral antibiotics; deep wound infection was defined as any infection within 1 year of injury which required intravenous antibiotics or surgical debridement in the operating room. Complications included (not all were found but the following were specifically searched) superficial infection (defined as cellulitis requiring oral antibiotics), deep infection (defined as requiring intravenous antibiotics or surgical debridement), urinary tract infection, pneumonia, pulmonary embolism, deep venous thrombosis, acute renal failure or insufficiency, nonunion, delayed union, compartment syndrome, osteomyelitis, nerve palsy, anoxic brain injury, cardiac ischemia or infarct, pancreatitis, or death.

**Results**: There was no increased risk for complication related to anemia itself (p=0.3). However, there was a significant risk for complication related to transfusion (p<0.01); furthermore, there was a dose-dependent effect with complication risk increasing with each unit transfused (p=0.02). Other factors such as age, injury severity score (ISS), and gender were considered and when adjusted did not change these results.

Conclusion: In young, healthy Orthopaedic trauma patients anemia does not appear to act as an independent risk factor for complications; however, allogeneic blood transfusion does appear to be a significant independent risk factor for complication and has a dose-dependent effect. Based on our findings from this retrospective study, we are designing a multi-specialty prospective study on Orthopaedic Trauma patients at our institution to determine if transfusion simply acts as a marker for patients at higher risk for complication due to injury or if transfusion might contribute directly to these complications.